CLINICAL TRIAL: NCT03775759
Title: Treatment of Tricuspid Valve Regurgitation in Patients Undergoing Left Ventricular Assist Device Implantation Study
Acronym: TVVAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Medtronic (Industry); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00072372
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Tricuspid Valve Insufficiency; Right Heart Failure; Heart Failure
Keywords: Left ventricular assist device; Tricuspid regurgitation; Right heart failure
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Failure | interventions — Replantation

STUDY DESIGN:
Intervention Model Description: Randomized controlled, non-blinded, single center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study arm (Experimental): Tricuspid valve ring annuloplasty or replacement at the time of LVAD implantation plus medical therapy
  Interventions: Procedure: Tricuspid valve repair or replacement
- Control arm (Active Comparator): LVAD implantation plus medical therapy
  Interventions: Other: Medical management of tricuspid regurgitation

INTERVENTIONS:
Procedure: Tricuspid valve repair or replacement — Available rings used at Duke include the Tri-Ad™ Adams Tricuspid Ring by Medtronic, the TAILOR™ FLEXIBLE ANNULOPLASTY RING by St. Jude Medical/Abbott, and the Carpentier-Edwards Physio II Ring by Edwards LifeSciences. Available valves used at Duke include the Mosaic™ Mitral Orbutrator by Medtronic, the Carpentier-Edwardes PERIMOUNT Magna Mitral Ease Pericardial Bioprosthesis by Edwards LifeSciences, the On-X Mitral Valve, by CryoLife, the Carbomedics Prosthetic Heart Valve by LivaNova, and the St. Jude Medical™ Mechanical Heart Valve by St. Jude Medical/Abbott.
  Arms: Study arm
Other: Medical management of tricuspid regurgitation — The medical therapy involved includes inotropic medications and diuretic medications, which are standard of care for patients in this population.
  Arms: Control arm

SUMMARY:
The purpose of this study is to determine the utility of tricuspid valve repair at the time of LVAD implantation for patients presenting with moderate or severe tricuspid regurgitation. The study will be a randomized trial for patients presenting for LVAD implantation to either tricuspid valve repair or no tricuspid valve repair. The data will be analyzed as both an intention to treat analysis as well as an "as treated" analysis with the primary outcome being rates of right ventricular dysfunction post LVAD implantation. Tricuspid valve repair for these patient is currently being done for some patients, without any strong data to either support such practice or negate it.

DETAILED DESCRIPTION:
This study is a prospective, single center, randomized trial. Up to 280 subjects will be enrolled.

Inclusion Criteria - Potential subjects must meet all inclusion criteria to participate.

* Planned LVAD implantation (either destination or bridge indication)
* 18 years of age or older
* Patients wilith mild tricuspid regurgitation (TR) during surgical planning will be screened for meeting inclusion criteria for this study.
* TR on pre-operative echo (within one week of procedure) (TTE or intraoperative TEE) quantified as moderate or severe with normal tricuspid valve leaflets

Exclusion Criteria

* Previous tricuspid valve surgery
* Previous LVAD
* Planned concurrent right ventricular assist device (RVAD) or extracorporeal membrane oxygenation (ECMO) at the time of LVAD operation or during the same hospitalization
* Preimplant RVAD or ECMO
* Planned thoracotomy approach for LVAD implantation
* Pregnant women

All subjects will undergo an intraoperative transesophageal echocardiogram (TEE) to evaluate their tricuspid valve. Subjects will be randomized in the operating room. Randomization will be stratified based on preoperative right ventricle dysfunction. Subjects will be randomized 1:1 to either of the following treatment arms:

* Study arm (Arm A) - Tricuspid valve ring annuloplasty or replacement at the time of LVAD implantation plus medical therapy
* Control arm (Arm B) - LVAD implantation plus medical therapy (the medical therapy involved includes inotropic medications and diuretic medications, which are standard of care for patients in this population)

Subjects will be monitored in the surgical and on the step down floor ICU, and follow-up data will be collected on subjects monthly from routine tests and clinic visits. This will include information on adverse events and any hospital readmissions, a quality of life questionnaire at their 6 and 12 month visit, and a six minute walk test at 3, 6, and 12 months. Cardiopulmonary exercise testing will be completed at 12 or greater months.

ELIGIBILITY:
Inclusion Criteria:

* Planned LVAD implantation (either destination or bridge indication)
* 18 years of age or older
* Patients will mild tricuspid regurgitation (TR) during surgical planning will be screened for meeting inclusion criteria for this study.
* Patients with moderate or graeter TR on pre-operative echo (within one week of procedure) (TTE or intraoperative TEE) will qualify for randomization

Exclusion Criteria:

* Previous tricuspid valve surgery
* Previous left ventricular assist device
* Planned concurrent right ventricular assist device (RVAD) or extracorporeal membrane oxygenation (ECMO) at the time of LVAD operation or during the same hospitalization
* Preimplant RVAD or ECMO
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients experiencing moderate or greater right heart failure within 6 months post-operatively | 6 months post-operatively
  Patients experiencing moderate or greater right heart failure as defined by Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) criteria
Proportion of patients experiencing moderate or greater right heart failure at 12 months post-operatively | 12 months post-operatively
  Patients experiencing moderate or greater right heart failure as defined by Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mendiola Pla M, Chiang Y, Nicoara A, Poehlein E, Green CL, Gross R, Bryner BS, Schroder JN, Daneshmand MA, Russell SD, DeVore AD, Patel CB, Katz JN, Milano CA, Bishawi M. Surgical Treatment of Tricuspid Valve Regurgitation in Patients Undergoing Left Ventricular Assist Device Implantation: Interim analysis of the TVVAD trial. J Thorac Cardiovasc Surg. 2024 May;167(5):1810-1820.e2. doi: 10.1016/j.jtcvs.2022.10.054. Epub 2022 Nov 16. PMID 36639288